CLINICAL TRIAL: NCT02910297
Title: The Pharmacokinetics of Cannabidiol (CBD) and Its Effects in Children With Severe Epilepsy
Status: Withdrawn | Type: Observational
Why Stopped: unable to recruit enough subjects on CBD
Sponsor: Gillette Children's Specialty Healthcare (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: CBD-PK-1
Record Dates: First submitted 2016-08-11; First posted 2016-09-22 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Dravet Syndrome; Lennox Gastaut Syndrome
Keywords: cannabidiol; Dravet Syndrome; Lennox Gastaut Syndrome
MeSH Terms: conditions — Epilepsies, Myoclonic; Lennox Gastaut Syndrome

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples collected to measure cannabidiol concentrations
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if cannabidiol (CBD) obtained via the state of Minnesota reduces seizures in patients with severe intractable epilepsy (Dravet Syndrome or Lennox Gastaut Syndrome), and to measure blood levels of CBD to help determine CBD concentration-response characteristics.

DETAILED DESCRIPTION:
Patients with medically refractory epilepsy who are registering to take CBD in the State of Minnesota will be offered the opportunity to participate in this study. If consent to participation is obtained, the patient (or more likely, the patient's guardian) will be asked to begin a seizure diary for at least a 7-day period prior (ideally, longer) to receiving the CBD, and to continue tracking seizures throughout the study. Upon receipt of CBD from the Minnesota dispensary, subjects will take their CBD as directed and will return to the clinic for a repeat visit (which is part of standard care) occurring 2-8 weeks after continual use of CBD. During these clinic visits, patients undergo blood draws to monitor their other prescribed AED concentrations as part of standard of care. In addition to the standard blood draw, the research participant will be asked to provide a blood sample of 5 ml to measure CBD concentrations. As most patients are instructed to take CBD two hours prior to their standard of care AEDs, clinical experience indicates that most patients are taking CBD quite early in the morning (around 6 AM). Thus, the time of sample collection will be recorded as hours post-dose, and will likely be nearer peak serum concentrations. If a study participant has an indwelling intravenous access port, they will be asked to provide an additional sample of 5 ml at least one hour after the initial sample. During the repeat visit, subjects will be asked to continue documenting seizure activity in their seizure diary while they continue their CBD treatment. Any changes to AEDs administered concurrently with CBD will also be recorded.

Subjects who are already on a stable regimen of CBD will also be eligible to participate. At a clinic visit, they will be asked to provide a blood sample of 5 ml, the time of each sample will be recorded as hours post-dose of CBD. They will also be asked to begin a seizure diary and continue tracking seizure activity. If a patient terminates their CBD treatment, they will be asked to continue tracking seizure activity after their last CBD dose until their follow-up clinic visit, to determine change in seizure activity while on and off CBD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Dravet Syndrome or Lennox-Gastaut Syndrome
* Patients who are planning to obtain medical cannabidiol
* Patients who are already taking medical cannabidiol and are planning to stop taking it.

Exclusion Criteria:

* Patients without a diagnosis of Dravet syndrome or Lennox-Gastaut syndrome

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects who have registered or plan to register with the state of Minnesota for taking medical cannabis and have severe intractable epilepsy (Dravet Syndrome or Lennox Gastaut Syndrome)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Reduction in seizures | a 7-day seizure diary completed at least twice within 3 months
  Subjects or parents/guardians of subjects will record seizure activity in seizure diaries both prior to and during cannabidiol administration

SECONDARY OUTCOMES:
Cannabidiol concentration | 1 time at a clinic visit within three months. If a patient has a port, they will be asked to provide an additional blood sample of 5 ml at least one hour after the first sample during the same clinic visit.
  Each subject will provide a blood sample of 5 ml to measure concentrations of cannabidiol

CONTACTS AND LOCATIONS:
Overall Officials: Samuel A Roiko, Ph.D., Principal Investigator — Gillette Children's Specialty Healthcare